CLINICAL TRIAL: NCT02981433
Title: Activation of the Sphingosine-1-phosphate (S1P) to S1P1 Receptor Subtype (S1PR1) Axis in Patients With Vulvodynia: Identification of Potential Relevant Biomarkers
Brief Title: Vulvodynia: Identification of Potential Relevant Biomarkers
Status: Completed | Type: Observational
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Cherie LeFevre, MD, Principal Investigator, St. Louis University
Other Study IDs: 27036
Record Dates: First submitted 2016-11-30; First posted 2016-12-05 (Estimated); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Vulvodynia
MeSH Terms: conditions — Vulvodynia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood leukocytes (PBLs) may provide a relevant biomarker to predict severity and pain induction outcomes as well as predict patient responses to anti-S1PR1 approaches.
Oversight: Data Monitoring Committee: No

SUMMARY:
Vulvodynia is a syndrome of unexplained vulvar pain that is frequently accompanied by physical disabilities, limitation of daily activities (such as sitting and walking), sexual dysfunction and psychologic disability. Originally suggested by McKay, the term "vulvodynia" has also been suggested by the International Society for the Study of Vulvar Disease Task Force to describe any vulvar pain. The incidence and prevalence of vulvodynia have not been well studied. Age distribution for the condition may range from the 20s to the 60s, and it is limited almost exclusively to white women. Obstetric and gynecologic history is usually unremarkable. Risk-taking sexual behavior is rare, and few patients have a history of sexually transmitted diseases. Vulvar pain usually has an acute onset, at times associated with episodes of vaginitis or certain therapeutic procedures of the vulva (cryotherapy or laser therapy). In most cases, vulvodynia becomes a chronic problem lasting months to years. Vulvar pain is frequently described as burning or stinging, or a feeling of rawness or irritation.

Most patients consult several physicians before being diagnosed. Many are treated with multiple topical or systemic medications, with minimal relief. In some cases, inappropriate therapy may even make the symptoms worse. Since physical findings are few and cultures and biopsies are frequently negative, patients may be told that the problem is primarily psychologic, thus invalidating their pain and adding to their distress.

DETAILED DESCRIPTION:
Sphingosine-1-phosphate (S1P) is a potent anti-apoptotic sphingolipid with potent pro-inflammatory actions which are driven in most part by activation of the S1P receptor subtype S1PR158. Biologically active S1P is generated by the phosphorylation of sphingosine, catalyzed by two sphingosine kinases (SphK1, SphK2). S1P levels are further regulated by its dephosphorylation by two phosphatases (SGPP1 and SGPP2) and through degradation by one lyase (SGPL1). Once released S1P initiates signaling through a family of five cognate G protein-coupled receptors (S1PR1-5), leading to various cellular responses9. S1P signaling has important roles in inflammation and cancer. S1P acting via the S1PR1 has been implicated in the development of pain of several etiologies as discovered by Salvemini and coworkers and subsequently extended by others. FTY720 (fingolimod/Gilenya®) is the first orally available agent approved by the FDA for the treatment of relapsing-remitting multiple sclerosis (MS). The work by Salvemini's group in providing a mechanistic basis for understanding chronic pain through the S1P/S1PR1 axis, provides a promising therapeutic target for the use of agents like FTY720 as a novel treatment for pain. Ongoing work by the Salvemini's lab suggests that increased expression of S1PR1 in circulating peripheral blood leukocytes (PBLs) may provide a relevant biomarker to predict severity and pain induction outcomes as well as predict patient responses to anti-S1PR1 approaches.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years of age
* Vulvar pain of at least 3 months' duration
* Localized (e.g. vestibulodynia, clitorodynia) or Generalized or Mixed
* Provoked or Spontaneous or Mixed Onset
* Temporal pattern

Exclusion Criteria:

* <18 or >70 years of age
* pregnant
* Not able to provide consent
* Patients with active vulvar dystrophies.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For patients with vulvodynia-related painwill be offered enrollment into the study. At their visit before treatment begins they will have:
  blood drawn ,(about 10ml-two teaspoons) this is research related. The ISSVD (The International Society for the Study of Vulvovaginal Disease) classification and diagnostic criteria for vulvodynia will be used for inclusion in this study.
  Vulvodynia - Vulvar pain of at least 3 months' duration,
  Descriptors:
  * Localized (e.g. vestibulodynia, clitorodynia) or Generalized or Mixed (localized and generalized)
  * Provoked (e.g. insertional, contact) or Spontaneous or Mixed (provoked and spontaneous)
  * Onset (primary or secondary)
  * Temporal pattern (intermittent, persistent, constant, immediate, delayed)
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
S1PR1 elevation | up to one year
  S1PR1 is elevated in the peripheral blood leukocytes (PBLs) of patients with vulvodyna-related pain.

CONTACTS AND LOCATIONS:
Overall Officials: Cherie LeFevre, MD, Principal Investigator — St. Louis University
Locations (2):
- United States (2):
  - St. Lukes Doctors South Office building, St Louis, Missouri
  - 1031 Bellevue office suite 200, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No